CLINICAL TRIAL: NCT07389889
Title: Percutaneous Robotic Navigation Microwave Ablation Versus CT-guided Microwave Ablation in the Treatment of Pulmonary Nodules With Ground-glass Opacity: A Prospective Randomized Controlled Trial
Brief Title: Percutaneous Robotic Navigation Microwave Ablation Versus CT-guided Microwave Ablation in the Treatment of Pulmonary Nodules With Ground-glass Opacity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: union TC1
Record Dates: First submitted 2025-12-10; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Nodules; Ground-glass Opacity
Keywords: ggo
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Experimental group: Microwave ablation under robot navigation (Active Comparator): Microwave ablation under robot navigation
  Interventions: Procedure: Robot
- Group B: CT-guided microwave ablation (Sham Comparator)
  Interventions: Procedure: CT scan

INTERVENTIONS:
Procedure: Robot — Microwave ablation guided by Robot or CT
  Arms: Group A: Experimental group: Microwave ablation under robot navigation
Procedure: CT scan — CT
  Arms: Group B: CT-guided microwave ablation

SUMMARY:
1. To compare the precision of robot-guided microwave ablation and CT-guided microwave ablation in the treatment of ground-glass nodules.
2. To evaluate the safety of robot-assisted microwave ablation and CT-guided microwave ablation in the treatment of ground-glass nodules.
3. Explore the application potential of robot navigation microwave ablation technology in the treatment of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 85 years
2. Nodules measuring 3-30mm with ground-glass opacities constituting ≥75% of the lesion
3. Preoperative clinical evaluation confirming no hilar or mediastinal lymph node metastasis and no distant metastasis
4. Patients diagnosed as stage IA primary peripheral lung cancer according to the UICC 8th TNM staging system, and with one of the following conditions:

   (i) cannot undergo surgical resection due to poor cardiopulmonary function or advanced age (ii) refusing or unwilling to undergo surgical resection (iii) with newly developed or residual pulmonary nodules after early-stage primary lung cancer surgery (iv) with unilateral lung disease who cannot undergo unilateral surgical resection (v)with multiple primary lung cancers unsuitable for surgical resection
5. Preoperative ECOG physical status score is 0/1
6. ASA score is I-III
7. Patients voluntarily participate in this study and sign the informed consent form

Exclusion Criteria:

1. Smoking cessation duration <2 weeks
2. Lesions adjacent to pulmonary artery-vein main trunks
3. Lesions near the hilum or adjacent to lobar bronchi
4. Pregnancy or lactation status
5. Severe mental disorders
6. History of other malignancies within 5 years
7. Unstable angina or myocardial infarction within 6 months with coronary angiography showing severe stenosis of major coronary branches
8. Cerebral infarction or hemorrhage within 6 months
9. Continuous systemic corticosteroid therapy within 1 month
10. Patients or their authorized persons who do not wish to comply with the study protocol
11. Patients with other investigator-assessed ineligibility for the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of puncture | 24 month
  The proportion of patients who are successfully punctured to the target pulmonary nodule on the first attempt of puncture among all patients; whether the puncture is successful is validated by CT scan.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol